CLINICAL TRIAL: NCT07374159
Title: Severe Mental Disorders, Chronicity and Sedentary Behaviour: Usability and Effectiveness of the "Sit Less, Move More" Program as an Integrated Service at Osonament
Brief Title: Sit Less, Move More Program as an Integrated Service at Osonament
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Universitària del Bages (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SMI25
Record Dates: First submitted 2025-12-05; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Sever Mental Illnes
Keywords: sever mental illness; physical activity; sedentary behaviour
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Sit less and move more
- Comparator (Active Comparator)
  Interventions: Other: Actual care

INTERVENTIONS:
Behavioral: Sit less and move more — The "Sit Less, Move More" program was implemented between February and May 2018, with a total duration of 16 weeks. The intervention was led by AG and delivered across three locations: the main Osonament center in Vic, the Estivill Camps center in Torelló, and the Mental Health Residential Home in Manlleu. Each participant received two weekly contacts: one face-to-face session and one telephone follow-up.
  During the face-to-face sessions, participants collaboratively selected walking routes and discussed strategies to increase daily activity at home. Educational materials and personal diaries were distributed to support self-monitoring and reflection. The telephone sessions served to reinforce behavioral agreements and encourage adherence to the weekly goals.
  Participants were grouped according to affinity and place of residence to facilitate autonomous group walks and improve accessibility and adherence.
  Arms: Intervention
Other: Actual care — The intervention involve normal or standarized healthcare delivered in Osonament center
  Arms: Comparator

SUMMARY:
People with severe mental illness (SMI), such as schizophrenia, bipolar disorder, or major depressive disorder, experience a life expectancy reduction of 10-20 years, largely due to chronic conditions like cardiovascular disease and type 2 diabetes. These individuals are less physically active and spend more time in sedentary behaviours (SB), which are associated with increased mortality, poor metabolic health, worse cognition, and lower quality of life. Traditional studies often rely on self-reported SB, which is unreliable, whereas objective measures like accelerometry provide more accurate data. Understanding SB patterns is essential for designing effective interventions to reduce prolonged sitting and improve health outcomes in this population.

This study aimed to describe daily SB patterns in outpatients with SMI and evaluate the feasibility of the "Sit Less, Move More" program integrated into routine care at Osonament, a community mental health center in Catalonia. The pragmatic intervention lasted 16 weeks and included two weekly contacts: face-to-face sessions for planning walking routes and strategies to increase activity, and telephone follow-ups to reinforce goals. Participants were grouped by affinity and residence to encourage autonomous walks, and the program was embedded within individual recovery plans. Ethical approval was obtained, and informed consent was secured.

Sedentary behaviour and physical activity were measured using the ActivPAL™ accelerometer, worn continuously for seven days at baseline and post-intervention. The device provided detailed data on sitting time, standing, light activity, and moderate-to-vigorous activity, as well as SB bouts categorized by duration. Self-perceived health was assessed using a visual analogue scale. From 412 potential candidates, 231 were invited, 60 enrolled, and 53 completed the program. Dropouts were due to psychiatric relapse, hospitalization, discharge, relocation, or loss of interest.

The study demonstrates the feasibility of integrating SB reduction strategies into community mental health services and highlights the importance of objective SB measurement. It provides a foundation for developing tailored interventions that break up prolonged sitting and promote movement among people with SMI, addressing a critical gap in improving physical health and reducing premature mortality in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Being an active user of Osonament
* Having a clinical diagnosis of a severe mental illness (e.g., schizophrenia, bipolar disorder, etc) in a stable plhase of the illness

Exclusion Criteria:

* Actively using toxics substances
* Had a predominant diagnosis other than a sever mental disorder
* Presented with medical contraindication that prevented safe participation in physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Physical activity levels | From enrollment to the end of intervention at 12 weeks
  Total physical activity levels will be measured though accelerometry using ActivPAL. Total levels of physical activity (light or moderate-high) will be recorded in minutes
Sedentary behaviour | From enrollment to the end of intervention at 12 weeks
  Patterns of sedentary behvaiour will be measured though accelerometry using ActivPAL. Patterns of sedentary behaviour will be recorded in minutes and bouts
Self-perceived health | From enrollment to th end of intervention at 12 weeks
  Self-perceived health was evaluated using a single-item visual analogue scale ranging from 0 to 100, where participants rated their general health status, with higher scores indicating better perceived health. This measure was chosen for its simplicity and feasibility in populations with severe mental disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundació Universitaria del Bages, Manresa, Barcelona, Spain